CLINICAL TRIAL: NCT00151957
Title: A Phase III, Multi-center, Open-label Study of Methylphenidate Transdermal System (MTS) in Pediatric Patients Aged 6-12 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Safety and Tolerability of SPD485 in Children Aged 6-12 Diagnosed With ADHD and Previously Participated in MTS Trials
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Collaborators: Noven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD485-303
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylphenidate transdermal system (Experimental): MTS Patch 27.5mg, 41.3mg, 55mg, and 82.5mg for 7 Weeks
  Interventions: Drug: Methylphenidate Transdermal System

INTERVENTIONS:
Drug: Methylphenidate Transdermal System — MTS Patch 27.5mg, 41.3mg, 55mg, and 82.5mg for 7 Weeks
  Other Names: MTS

SUMMARY:
This study will evaluate the long-term safety of MTS in the symptomatic treatment of children aged 6-12 diagnosed with ADHD

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a psychiatric disorder characterized by 3 main symptoms: inattention, hyperactivity and impulsivity. This study will evaluate the long-term safety of SPD485 in the symptomatic treatment of children aged 6-12 diagnosed with ADHD

ELIGIBILITY:
Inclusion Criteria:

* Subject must have participated in and completed SPD485-201 or participated in and completed a minimum of five of the seven weeks of double-blind treatment in study SPD485-302. Subjects who are participating in N17-021 may enroll in this study following completion of the End of Study/Termination visit procedures.
* Females of childbearing potential must have a negative urine pregnancy test at Baseline and must abstain from sexual activity that could result in pregnancy, or use acceptable contraceptives.

Exclusion Criteria:

* Subject was terminated from SPD485-102, SPD495-201, SPD485-302 OR N17-021 for non-compliance or experienced a serious adverse event resulting in termination from the antecedent protocols
* Female subject is pregnant or lactating

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2004-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events over 12 months. | Weekly

SECONDARY OUTCOMES:
ADHD-RS-IV scores | Weekly
Parent Global Assessment | Weekly
Clinical Global Impressions Scale | Weekly
Child's Sleep Habits Questionnaire | Weekly

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Findling RL, Wigal SB, Bukstein OG, Boellner SW, Abikoff HB, Turnbow JM, Civil R. Long-term tolerability of the methylphenidate transdermal system in pediatric attention-deficit/hyperactivity disorder: a multicenter, prospective, 12-month, open-label, uncontrolled, phase III extension of four clinical trials. Clin Ther. 2009 Aug;31(8):1844-55. doi: 10.1016/j.clinthera.2009.08.002. PMID 19808143